CLINICAL TRIAL: NCT05732948
Title: PD-1 Silent PSMA/PSCA Targeted CAR-T for the Treatment of Prostate Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Unicar-Therapy Bio-medicine Technology Co.,Ltd (Industry)
Collaborators: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCTPSMA-PSCA v1.0
Record Dates: First submitted 2018-08-05; First posted 2023-02-17 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- autologous T cells & cyclophosphamide (Experimental): This is a phase I dose escalation study to assess the safety and tolerability using increasing doses of engineered autologous T cells PD-1 silent targeted to PSMA/PSMA administered one day after pretreatment with cyclophosphamide.
  Interventions: Drug: autologous T cells & cyclophosphamide

INTERVENTIONS:
Drug: autologous T cells & cyclophosphamide — This is a phase I dose escalation study to assess the safety and tolerability using increasing doses of PD-1(programmed death 1)silent PSMA(prostate-specific membrane antigen)/PSCA(prostate stem cell antigen)targeted CAR-T administered one day after pretreatment with cyclophosphamide.

SUMMARY:
This is a phase I study which will test the safety of different doses of the patients own immune cells which have been changed to help recognize and destroy the cancer cells. The investigators want to find out what effects, good and/or bad, it has on the body and on the prostate cancer. The immune cells (T cells) used in this study will be the patients own immune cells. They will be removed from the patients blood, changed in the laboratory, and then put back into their body. T cells help the body fight infections. These cells may also kill cancer cells in some cases. Right now the patients T cells are unable to kill the cancer cells. For this reason, the physician will change the T cells by putting in a gene so that they may be able to better recognize and kill the prostate cancer cells. A gene is a portion of information which comes from the DNA and tells the cell what to do. This gene will be put into the patients T cells by a weakened virus. It is hoped that this approach will help the T cells recognize the prostate cancer tumor cells and possibly kill them. This is an entirely new treatment for prostate cancer and it is not known if it will have any beneficial or unexpected harmful effects.

DETAILED DESCRIPTION:
Immunotherapy has become the major breakthrough and the most promising treatment, with the host of development of tumor biology, molecular biology and immunology. It has become the fourth tumor treatment model after traditional tumor therapies (surgery, chemotherapy, radiotherapy) . With the development of the research field, the CAR-T cell basis and clinical research of various targets have achieved good results. PSCA, PSMA,RORγ are potential targets and spectacular paradigm in the diagnosis and treatment of prostate cancer. This study is for evaluation of the safety and efficacy of PD-1(programmed death 1)silent PSMA(prostate-specific membrane antigen)/PSCA(prostate stem cell antigen)targeted CAR-T for the Treatment of Castrate Metastatic Prostate Cancer

ELIGIBILITY:
Inclusion Criteria:

* Evidence of metastatic disease in bone on bone scan, CT scan, and/or by MRI atany time following the initial diagnosis of prostate cancer;
* The corresponding antigens such as PSMA and PSCA/PDL1 were highly expressed;
* Male patients aged between 18 and 65;
* Karnofsky score ≥ 60, ECOG≤ 2;
* Important organ function as defined by the following: cardiac ejection fraction ≥ 50%; electrocardiogram showed no obvious abnormalities; creatinine clearance rate calculated by using Cockcroft- Gault formula ≥40ml/min ; ALT/AST≤ 3×the institution normal upper limit; total bilirubin ≤2.0mg/dl; coagulation function: PT/ APPT<2 ×the institution normal upper limit; SpO2 >92%; Blood: hemoglobin>80g/L, ANC ≥ 1, PLT ≥ 50×109/L;
* There is measurable target lesion;
* Voluntary informed consent is given;

Exclusion Criteria:

* Immunosuppressive drugs or hormones were used a week before admission;
* Severe active infection;
* Human immunodeficiency virus (HIV) positive;
* Active hepatitis B or C infection;
* Past medical history of other malignancies. Not included: patients who have been cured at any time prior to the treatment of the skin basal or squamous cell carcinoma and cervical carcinoma in situ; the other tumor has not listed above, but has been used and only cured by surgery, without further treatment by other measures, the subjects of disease-free survival more than 5 years, can be included in the study;
* Patients participating in other clinical trials;
* The researchers thought the subjects were unfit for inclusion or unable to participate in or complete the study;
* Patients with congenital immunodeficiency;
* There is a history of myocardial infarction and serious arrhythmia within six months;

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2018-08-02 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Tumor response is assessmented with Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 | 8 weeks
  Dose escalation is based on the dose limiting toxicity (DLT). In this phase I trial, dose escalation will be based on the DLT, defined as a grade 3 or 4 toxicity (excluding alopecia, fatigue) developing after infusion of the T cells as graded by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events Scale (CTCAE) Version 3.0. Only toxicities that are possibly, probably, or definitely related to treatment will be considered DLTs. Patients will be observed for DLTs four weeks (28 days) from the T cell infusion

SECONDARY OUTCOMES:
Asverse event is evaluated with CTCAE, version 4.0 | 8 weeks
  1. Changes in bone metastases [ Time Frame: Week 12 then every 3 months ]
  2. Changes in biomarkers of bone metastasis and metabolism [ Time Frame: Week 4 and week 12 ]
  3. Changes in circulating tumor cells [ Time Frame: Weeks 4, 12, 24 and every 3 months ]
  4. Humoral and cell-mediated immunity to PSMA/PSCA and other known prostate cancer antigens [ Time Frame: Weeks 12 and 24 ]
  5. To assess patterns of change in PSA. [ Time Frame: 5 years ]
  6. To track the persistence, accumulation, and migration of genetically retargeted anti-PSMA/PSCA autologous T cells [ Time Frame: 2 years ]

CONTACTS AND LOCATIONS:
Overall Officials: Tang Xiaowen, Study Chair — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, China

IPD SHARING:
Plan to Share IPD: No